CLINICAL TRIAL: NCT00627211
Title: A Double-blinded, Randomized Trial Comparing Carbondioxide(CO2)and Air Insufflation in Oesophago-gastro-duodenoscopy (OGD)
Brief Title: Carbon Dioxide Versus Air Insufflation in Oesophago-gastro-duodenoscopy (OGD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Principal Investigator, Geir Hoff, Professor, Norwegian Department of Health and Social Affairs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STHF Gastro BS1
Record Dates: First submitted 2008-02-06; First posted 2008-02-29 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Pain
Keywords: quality assessment; pain reduction; gastroscopy; carbondioxide insufflation; Patient satisfaction
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Room air insufflation (No Intervention): Air used for insufflation during gastroscopy to expand the lumen for inspection of the mucosal lining. This is current standard procedure, i.e. no experimental intervention.
- CO2 insufflation (Experimental): CO2 used for insufflation during gastroscopy to expand the lumen for inspection of the mucosal lining. This is not standard procedure and therefore experimental intervention.
  Interventions: Procedure: CO2 insufflation

INTERVENTIONS:
Procedure: CO2 insufflation — From the CO2 rack through the endoscopy rack CO2 will be insufflated to visualize the mucosa during oesophagogastroduodenoscopy.
  Arms: CO2 insufflation

SUMMARY:
Comparison on the effect on patient pain and discomfort by using CO2 instead of air for insufflation during gastroscopy.

DETAILED DESCRIPTION:
To achieve a satisfactory examination of the GI tract it needs to be distended during endoscopic procedures. After the examinations many patients complain of abdominal pain and discomfort. This pain has been substantially reduced by substituting room air with CO2 in both colonoscopies and ERCPs. The use of CO2 during colonoscopy has become routine practice at many endoscopy centers.

In our study we will test the hypothesis that abdominal pain after gastroscopies also can be reduced by substituting room air with CO2.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for OGD at the outpatient clinic of Telemark Hospital

Exclusion Criteria:

* Age <18
* Inability to give an informed concent
* Unsatisfactory norwegian language skills
* Patients not willing to participate
* COPD with dyspnoea NYHA 3-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pain after OGD | 0-48 hours

SECONDARY OUTCOMES:
Pain during OGD | 24 hours